CLINICAL TRIAL: NCT07087990
Title: The Effect of Virtual Reality Glasses and Stress Ball on Anxiety, Pain, and Satisfaction in Patients Undergoing Coronary Angiography: A Randomized Controlled Study
Brief Title: Effect of VR Glasses and Stress Ball on Anxiety in Coronary Angiography Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Sabahattin Zaim University (Other)
Responsible Party: Principal Investigator, Rabia Ozdemir, Principal Investigator, Istanbul Sabahattin Zaim University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IZU-EC-2024-10
Record Dates: First submitted 2025-07-03; First posted 2025-07-28 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Coronary Angiography (CAG); Anxiety; Pain
Keywords: Coronary Angiography; Virtual Reality; Stress Balls; Anxiety; pain; Satisfaction Levels
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: randomize kontrollü
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VR Group"Participants in this group were provided with virtual reality glasses during coronary angio (Experimental): Participants in this group were provided with virtual reality glasses during coronary angiography to assess the effect on anxiety, pain, and satisfaction.
  Interventions: Device: Virtual Reality Glasses
- Stress Ball Group (Experimental): Participants in this group used a stress ball during coronary angiography to evaluate its effect on anxiety, pain, and satisfaction.
  Interventions: Other: Stress Ball
- Control Group (No Intervention): Participants in this group received standard care during coronary angiography without the use of virtual reality glasses or stress ball. Anxiety, pain, and satisfaction levels were assessed

INTERVENTIONS:
Device: Virtual Reality Glasses — articipants in the VR group used virtual reality glasses during coronary angiography to reduce anxiety and pain and improve satisfaction.
  Arms: VR Group"Participants in this group were provided with virtual reality glasses during coronary angio
Other: Stress Ball — articipants in the stress ball group used a stress ball during coronary angiography to evaluate its effects on anxiety, pain, and satisfaction.
  Arms: Stress Ball Group

SUMMARY:
This randomized controlled trial aimed to evaluate the effects of virtual reality (VR) glasses and the use of a stress ball on anxiety, pain, and satisfaction levels in patients undergoing coronary angiography. Participants were randomly assigned to three groups: one group received both VR and stress ball interventions during the procedure, while the control group received standard care. Anxiety, pain, and satisfaction levels were assessed and compared across the three groups at the conclusion of the procedure. The study seeks to contribute to evidence on non-pharmacological methods to improve patient comfort during invasive cardiac procedures.

DETAILED DESCRIPTION:
This randomized controlled trial aimed to evaluate the effects of virtual reality (VR) glasses and the use of a stress ball on anxiety, pain, and satisfaction levels in patients undergoing coronary angiography. Participants were randomly assigned to three groups: one group received both VR and stress ball interventions during the procedure, while the control group received standard care. Anxiety, pain, and satisfaction levels were assessed and compared across the three groups at the conclusion of the procedure. The study seeks to contribute to evidence on non-pharmacological methods to improve patient comfort during invasive cardiac procedures.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation in the study
* Age 18 years or older
* Undergoing coronary angiography for the first time
* Cognitive ability to answer the questions
* No diagnosis of anxiety disorder and no use of medication for anxiety / no psychiatric diagnosis
* No physical disability preventing the use of the stress ball
* No problems with vision, hearing, or understanding

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Change in State Anxiety Inventory (SAI) Scores | Before and immediately after coronary angiography procedure
  the study will measure changes in situational anxiety levels of patients undergoing coronary angiography, using the State Anxiety Inventory (SAI) before and after the procedure with virtual reality glasses and stress balls. The SAI consists of 20 items rated on a 4-point Likert scale, with total scores ranging from 20 to 80; higher scores indicate higher anxiety.

SECONDARY OUTCOMES:
Change in Anxiety Visual Analogue Scale (VAS) Scores | Before and immediately after coronary angiography procedure
  Patients' anxiety levels will be assessed before and after coronary angiography using a 10 cm Visual Analogue Scale (VAS), where 0 indicates no anxiety and 10 indicates extreme anxiety.
Change in Pain Visual Analogue Scale (VAS) Scores | Before and immediately after coronary angiography procedure
  Patients' pain levels will be evaluated before and after coronary angiography using a 10 cm Visual Analogue Scale (VAS), where 0 means no pain and 10 indicates worst possible pain.

OTHER OUTCOMES:
Satisfaction with Virtual Reality Glasses Application | Immediately after virtual reality glasses intervention
  Patient satisfaction will be assessed using a 4-item custom form developed specifically for this study. The first item uses a 0 to 10 Visual Analogue Scale (VAS), where 0 indicates "not satisfied at all" and 10 indicates "extremely satisfied". The remaining items assess patient preferences and recommendations using multiple-choice questions (yes/no/undecided). Higher VAS scores reflect greater satisfaction.
Satisfaction with Stress Ball Application | Immediately after stress ball intervention
  Patient satisfaction will be evaluated using a 4-item form developed for this study. The first item uses a 0 to 10 Visual Analogue Scale (VAS), where 0 indicates no satisfaction and 10 indicates the highest satisfaction. The remaining three items gather feedback through multiple-choice responses. Higher VAS scores indicate greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Zülfünaz Özer, PhD, Study Chair — İstanbul Sabahattin Zaim University
Locations (1):
- Istanbul Sabattin Zaim Üniversitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
At this time, individual participant data (IPD) will not be shared due to concerns about patient privacy and confidentiality. Additionally, data sharing procedures are still under development. We are committed to protecting participants' personal information in accordance with applicable regulations and institutional policies.